CLINICAL TRIAL: NCT03247634
Title: Getting Ahead for Cancer Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CASE11Z17
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Cancer Prevention
Keywords: getting ahead; vulnerable population; safety net practice network

STUDY DESIGN:
Intervention Model Description: Interrupted Time Series - All cohorts will receive the Getting Ahead program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Getting Ahead Program (Experimental): 12 staggered cohorts will be given the Getting Ahead program, using the established Getting Ahead in a Just-Gettin'-By World program. Six practices will be used. Each participant will come in for 16 session over an eight week period and will be followed up six months post intervention
  Interventions: Behavioral: Getting Ahead in a Just-Gettin'-By World

INTERVENTIONS:
Behavioral: Getting Ahead in a Just-Gettin'-By World — The Getting Ahead program is a unique welldeveloped program that allows carefully guided introspection toward the crafting of tailored solutions aimed at addressing complex social determinants of health among individuals living in vulnerable populations where the achievement of health equity often seems unattainable. The important lens of health equity is a key component of this proposal and is consistent with the American Cancer Society overarching emphasis on reduction of health disparities and achievement of health equity.

SUMMARY:
A new, practical program, entitled Getting Ahead in a Just-Gettin'-By World, provides a novel approach to addressing this previously intractable problem. During the progression through the Getting Ahead program, individuals develop an understanding of the hidden rules of economic class and have an opportunity to craft a hopeful future story based on the practical concepts investigated in the modules. Getting Ahead has shown great success in various organizations and communities in multiple sectors, including healthcare, but has not been studied in the context of advancing cancer prevention and control.

DETAILED DESCRIPTION:
The study team hypothesizes that the Getting Ahead program, applied in safety net practices with primary care patients living in poverty, will improve cancer prevention and early detection activities, mediated by a shift in future orientation gained through the program.

This pilot study aims to adapt, apply, and evaluate the established Getting Ahead program in a health care setting and assess its effect on cancer prevention and early detection activities for vulnerable populations. By generating process and outcome data on a novel intervention to help people advance out of poverty, this research will set the stage for larger intervention studies, and also will advance understanding of the mechanisms by which growing a future orientation can improve cancer preventive service delivery among vulnerable populations.

Specifically, this study aims to:

1. Implement Getting Ahead among cohorts of patients at a network of safety net practices.
2. Assess the paradigm shift in developing a future orientation associated with participation in the Getting Ahead program.
3. Evaluate the effect of the Getting Ahead program and its associated paradigm shift on graduates' cancer prevention and early detection activities.

ELIGIBILITY:
Inclusion Criteria:

* Interest and willingness to commit to the 8 week Getting Ahead training program that will occur over 16 sessions occurring twice a week
* Willingness to commit to follow-up with his/her primary care provider after completion of the Getting Ahead training program
* Willingness to be randomized to an immediate or delayed (by 8 weeks) start date
* Ability to speak English

Exclusion Criteria:

* There are no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Change in composite score of cancer prevention | From baseline up to 3 years
  Change in composite score of cancer prevention based on changes in cognition, intention and behavior regarding tobacco reduction, fruit and vegetable consumption, and physical activity; Immunizations for human papillomavirus (HPV) or hepatitis B; Age/sex appropriate use of Pap tests, mammograms, stool tests, endoscopy or imaging studies for colorectal cancer

SECONDARY OUTCOMES:
Change in composite score of progress toward a future orientation | From baseline up to 3 years
  change in composite scores based on 11 resource areas with a score ranging from 1-5 (total scores ranging from 11-55 with 55 being the most stable score). The score indicates the level of stability

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Gullett, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States